CLINICAL TRIAL: NCT06206681
Title: Efficacy and Safety of Ultrapulse Carbon Dioxide Laser Treatment in Eyelid Tumors
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yingfeng Zheng, Principal Investigator, Sun Yat-sen University
Other Study IDs: 2023KYPJ286
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Eyelid Tumor; Xanthelasma Palpebrarum; Pigmented Nevi; Keratosis
MeSH Terms: conditions — Eyelid Neoplasms; Xanthomatosis; Nevus, Pigmented; Keratosis | interventions — Lasers, Gas

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ultrapulse Carbon Dioxide Laser: The study investigates the use of the Ultrapulse Carbon Dioxide Laser for the excision of eyelid lesions, including xanthelasma, pigmented nevi, keratoses, and so on.
  Interventions: Procedure: Ultra-pulsed Carbon Dioxide Laser

INTERVENTIONS:
Procedure: Ultra-pulsed Carbon Dioxide Laser — Excision of eyelid lesion
  Other Names: CO2 Laser

SUMMARY:
This study aims to assess the long-term efficacy and safety of ultrapulse carbon dioxide (CO₂) laser excision in the treatment of eyelid tumors, including xanthelasma, pigmented nevi, keratoses, and so on.

DETAILED DESCRIPTION:
-Background: The assessment of the efficacy and safety of Ultrapulse CO₂ laser in treating eyelid lesions is crucial for clinical applications. This study aims to evaluate the effectiveness of super-pulsed CO₂ laser in treating different types of eyelid lesions, particularly marginal and large lesions, to provide comprehensive clinical guidance and decision support.

-Main Objectives: A retrospective analysis of the efficacy and safety of Ultrapulse CO₂ laser treatment for various types of eyelid lesions, including xanthelasma, pigmented nevi, keratoses, and so on.

-Study Design: This study will include 1000 patients diagnosed with eyelid lesions, including xanthelasma, pigmented nevi, keratoses, and so on. All patients undergoing Ultrapulse CO₂ laser treatment. The evaluation will focus on the efficacy and safety of Ultrapulse CO₂ laser treatment for different types of eyelid lesions.

-Study Population and Anticipated Enrollment: Patients with eyelid lesions (n=1000)

-Inclusion Criteria: Clinically diagnosed with eyelid lesions, including xanthelasma, pigmented nevi, keratoses, and so on.

No history of photosensitivity, bleeding, or coagulation disorders Willing to attend follow-up appointments as scheduled

-Exclusion Criteria: Presence of infection in the target area Allergy to lidocaine Keloid-prone or poor skin repair ability Pregnant or lactating Recent history of severe infectious diseases, active skin diseases, or major diseases affecting the cardiovascular, liver, kidney, endocrine, and hematopoietic systems History of malignant tumors or immune system disorders

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with eyelid lesions, including xanthelasma, pigmented nevi, keratoses, and so on.
* No history of photosensitivity, bleeding, or coagulation disorders
* Willing to attend follow-up appointments as scheduled

Exclusion Criteria:

* Presence of infection in the target area
* Allergy to lidocaine
* Keloid-prone or poor skin repair ability
* Pregnant or lactating
* Recent history of severe infectious diseases, active skin diseases, or major diseases affecting the cardiovascular, liver, kidney, endocrine, and hematopoietic systems
* History of malignant tumors or immune system disorders

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A cohort of 1000 patients with eyelid tumors, including various types of tumors. Inclusive of xanthelasma, pigmented nevi, keratoses, and so on.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Clearance rate | 12 months
  The lesion clearance rate was classified as the proportion of the lesion cleared (<50%; 50-75%; 76-99%; or >99%).
Recurrence rate | 12 months
  Recurrence was defined as the regrowth of a new xanthelasma lesion within the previously excised area.

SECONDARY OUTCOMES:
Postoperative complications | 12 months
  Lesion recurred, minor trichiasis, partial sparse to absent eyelashes, hypertrophic scar, hyperpigmentation
Investigator's Global Assessment (IGA) score | 12 months
  Investigator's Global Assessment (IGA) score for measuring improvement in clinical outcomes: 1=worsened; 2=no change; 3=minor improvement; 4=moderate improvement; 5=marked improvement; 6=near-total improvement; and 7=total improvement.
Patient satisfaction score | 12 months
  Patient satisfaction was evaluated subjectively by the physician on a f ve-point scale, as follows: 0=no change; 1=minor improvement; 2=moderate improvement; 3=marked improvement; 4=near-total or total improvement.
Number of treatment sessions | 12 months
  Number of treatment sessions for complete clearance

CONTACTS AND LOCATIONS:
Overall Officials: Xianchai Lin, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Sun Yat-sen University, Guanzhou, China

IPD SHARING:
Plan to Share IPD: No